CLINICAL TRIAL: NCT00234481
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL844 Administered Orally to Subjects With Chronic Lymphocytic Leukemia
Brief Title: Safety Study of XL844 in Subjects With Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to slow enrollment
Sponsor: Exelixis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL844-001
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Drug: XL844

SUMMARY:
The purpose of this study is to assess the safety and tolerability of different doses of XL844 when given orally to adults with recurrent or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent or refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL)
* Prior treatment with at least 2 systemic chemotherapy regimens for CLL
* Life expectancy of >3 months
* Adequate liver and kidney function
* Absolute neutrophil count ≥500/mm3; platelets ≥50,000/dL; hemoglobin ≥9 g/dL
* Willing to use accepted method of contraception during the course of the study
* Negative pregnancy test (females)
* Written informed consent

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4-6 weeks of the start of treatment (depending on the therapy)
* Investigational drug within 30 days of the start of treatment
* Uncontrolled intercurrent illness such as infection or cardiovascular disease
* Pregnant or breastfeeding women
* Subjects known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - City of Hope National Cancer Center, Duarte, California
  - UCSD Moores Cancer Center, San Diego, California
  - UT MD Anderson Cancer Center, Houston, Texas